CLINICAL TRIAL: NCT00189566
Title: National, Randomized, Phase II Study Comparing Efficacy of Weekly Administration of Paclitaxel in Monotherapy or in Combination With Topotecan or Carboplatin in Patients With Epithelial Ovarian Cancer in Early Relapse
Brief Title: Taxol® in Monotherapy or in Combination With Topotecan or Carboplatin in Patients With Epithelial Ovarian Cancer in Early Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAR\TAXHY
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Malignant Tumor of Peritoneum
Keywords: Relapse within 6 months; Previously received taxane derivative
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Paclitaxel; Topotecan; Carboplatin

INTERVENTIONS:
Drug: Paclitaxel
Drug: Topotecan
Drug: Carboplatin

SUMMARY:
This study will look at the efficacy and safety of weekly administration of paclitaxel (Taxol®) in monotherapy compared to paclitaxel in combination with topotecan or carboplatin in patients with ovarian cancer in early relapse.

DETAILED DESCRIPTION:
The main purpose of this research study is to find out if treatment of early relapse of ovarian or fallopian tube or peritoneal cancer with paclitaxel (Taxol*) weekly administered, in lower doses in combination with topotecan (Hycamtin*) or carboplatin will improve efficacy compared to weekly administration of paclitaxel in monotherapy. Tolerance in the three groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18
* Histologically proven diagnosis of cancer of the ovary, the fallopian tube or peritoneum
* Peritoneal and/or nodes and/or visceral metastases
* Disease in progression under treatment or within 6 months after a first or second platinum-based line
* A period of 3 weeks between last chemotherapy and inclusion
* Measurable disease (Response Evaluation Criteria in Solid Tumors [RECIST] criteria) or cancer antigen (CA) 125 assessable disease (Gynecologic Cancer Intergroup [GCIG] criteria)
* ECOG performance status < 2
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Previously received weekly administration of paclitaxel chemotherapy
* Involved in a trial within the last 30 days
* Previously received a bone marrow autogreffe or irradiation of the abdomen within 5 years, due to intensive chemotherapy
* Prior diagnosis of malignancy
* History of ischemic cardiopathy, congestive heart failure (New York Heart Association [NYHA] > 2), arrhythmia, hypertension, or significant valvulopathy
* Pre-existing motor or sensory neurologic pathology or symptoms National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) grade > 2
* Bone marrow, renal, or hepatic insufficiency
* Severe active infection or occlusive or sub-occlusive disease
* History of symptomatic brain metastases
* Fertile women not using adequate contraceptive methods
* Pregnant or breast feeding women
* Hypersensitivity to compounds chemically related to paclitaxel, topotecan, or carboplatin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2004-04; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of patients in the three groups

SECONDARY OUTCOMES:
Overall survival
Rate of response and rate of progression at the end of treatment
Qualitative and quantitative toxicities
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Laure Chauvenet, MD, PhD, Study Director — Hôpital Hôtel Dieu
Locations (1):
- Hôpital Hotel Dieu, Paris, France